CLINICAL TRIAL: NCT02895828
Title: Clinical Practice Guideline With Core Stabilization and Strengthening Exercise Programs for Low Back Pain With Clinical Lumbar Instability
Brief Title: Effects of Core Stabilization and Strengthening Exercise on Quality of Life in Clinical Lumbar Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Wantanee Yodchaisarn, Principal investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE562257
Record Dates: First submitted 2014-11-24; First posted 2016-09-12 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core Stabilization Exercise (CSE) (Experimental): The participants asked to performed CSE program, 20 min/session, 2 session/week, 10 weeks
  Interventions: Other: Core Stabilization Exercise
- General Strengthening Exercise (GSE) (Experimental): The participants asked to performed GSE program, 20 min/session, 2 session/week, 10 weeks.
  Interventions: Other: General Strengthening Exercise

INTERVENTIONS:
Other: Core Stabilization Exercise — the participants asked to performed CSE program, 20 min/session, 2 session/week, 10 weeks
  Arms: Core Stabilization Exercise (CSE)
Other: General Strengthening Exercise — the participants asked to performed GSE program, 20 min/session, 2 session/week, 10 weeks
  Arms: General Strengthening Exercise (GSE)

SUMMARY:
This study will compare the effects of 2 exercise programs including core stabilization exercise and general trunk strengthening exercise programs on trunk muscle activity, physical dysfunction, quality of life and lumbar motion in low back pain patient with clinical lumbar instability.

DETAILED DESCRIPTION:
Clinical lumbar instability is the one of causes of chronic low back pain, that affects to pain intensity and quality of life. For clinical studies using core stabilization exercise (CSE) as treatment have revealed conflicting findings on pain, functional disability and muscle responses in chronic low back pain. The CSE promotes local muscle system that to provide lumbar stability. However, the stability of spine related to global muscle system, that using in this study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain due to clinical lumbar instability

Exclusion Criteria:

* Specific low back pain
* Cuada equine syndrome
* Neurological deficit

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Effect of 2-exercise on quality of life | Change from baseline at 10-week after training session, and follow up session
  health-related quality of life was measured by using SF-36 questionnaire

SECONDARY OUTCOMES:
Effect of 2-exercise on physical disability | Change from baseline at 10-week after training session, and follow up session
  Physical disability was measured by using Oswestry disability index
Effect of 2-exercise on trunk muscle activity | Change from baseline at 10-week after training session, and follow up session
  Trunk muscle activity was measured by using surface EMG
Effect of 2-exercise on lumbar segmental motion | Change from baseline at 10-week after training session, and follow up session
  Lumbar segmental motion was measured by using radiography
Effect of 2-exercise on pain intensity | Change from baseline at 10-week after training session, and follow up session
  Pain intensity was measured by using numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Wantanee Yodchaisarn, M.Sc., Principal Investigator — The Research Center in Back, Neck, Other Joint Pain and Human Performance (BNOJPH), Khon Kaen University, Thailand
Locations (1):
- Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen, Thailand

REFERENCES:
- [Background] Puntumetakul R, Areeudomwong P, Emasithi A, Yamauchi J. Effect of 10-week core stabilization exercise training and detraining on pain-related outcomes in patients with clinical lumbar instability. Patient Prefer Adherence. 2013 Nov 19;7:1189-99. doi: 10.2147/PPA.S50436. eCollection 2013. PMID 24399870
- [Background] Javadian Y, Behtash H, Akbari M, Taghipour-Darzi M, Zekavat H. The effects of stabilizing exercises on pain and disability of patients with lumbar segmental instability. J Back Musculoskelet Rehabil. 2012;25(3):149-55. doi: 10.3233/BMR-2012-0321. PMID 22935853